CLINICAL TRIAL: NCT04485221
Title: A Natural History Study in Children With a TECPR2 Mutation
Brief Title: TECPR2 Observational Study
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202001737
Record Dates: First submitted 2020-06-18; First posted 2020-07-24 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: TECPR2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood and
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with a TECPR2 mutation: Children with a TECPR2 mutation, age 18 months to 12 years old.
  Assessments will include collection of genetic mutation reports, functional assessments, and questionnaires. There will be a singular blood draw and skin biopsy.

SUMMARY:
The purpose of this study is to learn more about the disease progression in patients with a TECPR2 mutation.

DETAILED DESCRIPTION:
A mutation in the tectonin beta-propeller repeat containing 2 (TECPR2) gene can disrupt the cellular process of autophagy resulting in neuronal cell death. This disruption leads to a form of spastic paraplegia with the additional disruption to involuntary body processes, such as respiration and thermoregulation. This study will provide valuable information about the natural progression of children with a TECPR2 mutation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (and assent where appropriate) before any study procedures take place;
* Male or female;
* 18 months to 12 years old, at enrollment; and
* Have a diagnosis of TECPR2-Related disorder, as defined by biochemical criteria AND/OR genetic mutation analysis, AND demonstrate clinical findings such as autophagy, developmental delay, hypotonia, or other positive findings.

Exclusion Criteria:

* Subject is unable to comply with study requirements; or
* Have any other concurrent condition that, in the opinion of the investigator, would make the subject unsuitable for the study.

Ages: 18 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with TECPR2-Related disorder, confirmed by genetic mutation analysis and demonstrates clinical findings such as autophagy, developmental delay, hypotonia, or other positive findings.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
Disease progression | Baseline up to 24 months
  This will be monitored through medical history, physical exams, and a neurological exam.

SECONDARY OUTCOMES:
Functional assessment: Gross Motor Function Measure | Baseline up to 24 months
  This evaluative measure of motor function is designed for quantifying change in the gross motor abilities of children.
Functional assessment: Gross Motor Function Classification System | Baseline up to 24 months
  This measures the functional level of the patient based on their age.
Functional assessment: Timed Tests | Baseline up to 24 months
  Timed tests for ambulant children will include time to run 10 meters, time to climb four stairs, and time to rise from the floor from supine.
Functional assessment: Muscular Strength Testing | Baseline up to 24 months
  Muscle strength will be assessed for grip, pinch, quadriceps, hamstrings, biceps, and triceps.
Functional assessment: Ankle Dorsiflexion Range of Motion | Baseline up to 24 months
  This measurement is used to evaluate the degree of ankle contracture in a participant.
Patient Reported Outcomes: Pediatric Quality of Life Inventory | Baseline up to 24 months
  A questionnaire used for measuring health-related quality of life in healthy children and adolescents and those with acute and chronic illnesses.
Patient Reported Outcomes: Pediatric Evaluation of Disability Inventory Computer Adaptive Test | Baseline up to 24 months
  This questionnaire measures the extent to which the caregiver or child takes responsibility for managing complex, multi-step life tasks.

CONTACTS AND LOCATIONS:
Locations (1):
- Jenna Lammers, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oz-Levi D, Gelman A, Elazar Z, Lancet D. TECPR2: a new autophagy link for neurodegeneration. Autophagy. 2013 May;9(5):801-2. doi: 10.4161/auto.23961. Epub 2013 Feb 25. PMID 23439247
- [Background] Oz-Levi D, Ben-Zeev B, Ruzzo EK, Hitomi Y, Gelman A, Pelak K, Anikster Y, Reznik-Wolf H, Bar-Joseph I, Olender T, Alkelai A, Weiss M, Ben-Asher E, Ge D, Shianna KV, Elazar Z, Goldstein DB, Pras E, Lancet D. Mutation in TECPR2 reveals a role for autophagy in hereditary spastic paraparesis. Am J Hum Genet. 2012 Dec 7;91(6):1065-72. doi: 10.1016/j.ajhg.2012.09.015. Epub 2012 Nov 21. PMID 23176824
- See also: Genetic home reference for TECPR2 — https://ghr.nlm.nih.gov/gene/TECPR2#normalfunction